CLINICAL TRIAL: NCT03205176
Title: A Phase I, Multicenter Dose-Escalation Study to Assess the Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of AZD5153 in Patients With Relapsed/Refractory Malignant Solid Tumors, Including Lymphomas
Brief Title: AZD5153 in Patients With Relapsed or Refractory Solid Tumors, Including Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6520C00001; REFMAL 495 (Other: Sarah Cannon Development Innovations, LLC)
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Malignant Solid Tumors; Lymphoma; Ovarian Cancer; Breast Cancer; Pancreatic Cancer; Prostate Cancer
Keywords: AZD5153; Olaparib; Malignant solid tumors; Lymphoma; Ovarian Cancer; BRD4; Triple negative breast cancer; Pancreatic cancer; Prostate cancer
MeSH Terms: conditions — Lymphoma; Ovarian Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Triple Negative Breast Neoplasms | interventions — AZD5153; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD5153 Monotherapy (Experimental): Patients will be enrolled in cohorts of up to 6 patients each in a dose escalating scheme to determine maximum tolerated dose (MTD). AZD5153 will be taken once per day (QD) or two times per day (BID) for 21 days as an oral capsule. Once the MTD is finalized, patients may be enrolled into an expansion cohort at the MTD.
  Interventions: Drug: AZD5153
- AZD5153 + Olaparib Combination Therapy (Experimental): Patients will be enrolled in cohorts of up to 6 patients each in a dose escalating scheme to determine MTD. AZD5153 will be taken as oral capsules BID in combination with 300 mg olaparib BID for 21 days.
  Interventions: Drug: AZD5153; Drug: Olaparib

INTERVENTIONS:
Drug: AZD5153 — AZD5153 is to be taken as oral capsules once or twice per day each day in 21 day cycles. Dosing will continue until disease progression or other study discontinuation criteria are met.
Drug: Olaparib — Olaparib, 300 mg, will be taken BID as oral capsules.
  Other Names: Lynparza
  Arms: AZD5153 + Olaparib Combination Therapy

SUMMARY:
This is a first-time-in-man (FTIM) multicenter, dose escalation study designed to investigate the safety, pharmacokinetics, and pharmacodynamics of AZD5153 in patients with malignant solid tumors, including lymphomas.

DETAILED DESCRIPTION:
The trial will be conducted in two parts, dose escalation and dose expansion. AZD5153 will be investigated as a monotherapy and in combination with olaparib.

AZD5153 monotherapy (dose escalation):

This part of the study will enroll patients with advanced solid malignancies, including lymphoma, and test safety and tolerability of AZD5153 administered as a monotherapy. The dose escalation will proceed by two-fold increments or through lower doses suggested by the CRM until an MTD as defined by dose-limiting toxicity is reached.

Single daily (QD) and twice daily (BID) dosing schedules will be explored in the monotherapy cohort. Additional dose levels or dosing schedules may be evaluated and recommended by study Safety Review Committee (SRC) based on the emerging PK and safety data.

When the AZD5153 monotherapy MTD is established, an expansion cohort consisting of up to 12 additional evaluable patients may be enrolled to confirm the safety and tolerability of the MTD. The dose expansion will be initiated and will enroll patients with histologically or cytologically confirmed platinum resistant or platinum-refractory high grade serous ovarian (HGSO) cancer.

Mandatory tumor biopsies at screening for ovarian cancer patients will be required for patient enrollment in the MTD dose expansion cohort. Optional on-treatment biopsies will be requested from consenting patients in the ovarian expansion cohort.

AZD5153 + olaparib combination:

Dose escalation of AZD5153 in combination with olaparib will also be investigated while the AZD5153 monotherapy dose escalation is ongoing and prior to determination of a monotherapy MTD.

The starting dose of AZD5153 in combination with olaparib will be a dose that has been shown to be safe and tolerated in monotherapy and has been chosen because clinical exposure achieved at this dose is equivalent to preclinical exposure causing tumour growth inhibition in animal models. If the starting dose in combination with olaparib is safe and tolerated, the dose of AZD5153 will be escalated, using the same method as for the monotherapy part of the study, keeping the olaparib dose fixed at 300 mg BID. Intermittent schedules as well as continuous BID or QD dosing of AZD5153 in combination with 300 mg BID olaparib might be tested until a safe and tolerated combination dose and schedule is determined. However, the total dose per cycle of AZD5153 used in combination with olaparib won't exceed the total dose per cycle that has been shown to be safe and tolerated as a monotherapy, and won't be higher than the dose declared to be the monotherapy MTD. If intermittent dosing is explored then the CRM will consider cumulative dosing rather than daily dosing.

AZD5153 and olaparib will be administered in continuous cycles of 21 days. The combination dose escalation part will run in parallel with the AZD5153 monotherapy part (dose escalation and expansion) and will continue until a safe and tolerated combination dose of the two agents is declared. Mandatory paired tumor biopsies at screening and on-treatment will be required for patients enrolled into the combination dose escalation.

Once a dose and schedule of AZD5153 in combination with olaparib is established, up to 12 additional evaluable patients might be enrolled to confirm the safety and tolerability of the dose and schedule of AZD5153 and olaparib in one or more of the indications where clinical activity is observed. Patients with platinum-resistant or platinum-refractory HGSO cancer, triple negative breast cancer, metastatic castration resistant prostate cancer, or pancreatic ductal adenocarcinoma will be eligible for the expansion cohort.

ELIGIBILITY:
Inclusion Criteria for all Patients:

1. Patient must be able to understand the nature of the study and provide a signed and dated, written informed consent prior to any study specific procedures, sampling or analyses.
2. Patients should have the ability and willingness to comply with the study and follow-up procedures.
3. Patients must have a solid tumor that is refractory to or intolerant of existing therapies known to provide clinical benefit for their clinical condition.
4. Age ≥ 18
5. Adequate organ function, determined by:

   * Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L
   * Platelets ≥ 100 X 10^9/L
   * Hemoglobin ≥ 9 g/dL
   * aPTT ≤1.5 x ULN
   * Total bilirubin ≤ 1.5 mg/dL
   * ALT and AST ≤ 2.5 x ULN if no liver involvement or ≤ 5 x ULN with liver involvement
   * Creatinine <1.5 times ULN concurrent with creatinine clearance >50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
6. Normotensive or well controlled blood pressure (BP) (<140/90), with or without current antihypertensive treatment. If there is a diagnosis or history of hypertension, patient must have adequately controlled BP on a maximum of 2 antihypertensive medications, as demonstrated by 2 BP measurements taken in the clinical setting by a medical professional within 1 week prior to enrollment. It is strongly recommended that patients who are on antihypertensive medications be followed by a cardiologist or a primary care physician for management of BP while on the study. Patients on a hypertensive medication must be willing and able to check and record twice daily BP readings for a minimum of 3 weeks.
7. ECOG performance status of 0-1
8. Life expectancy ≥ 3 months
9. Ejection fraction (EF) > 50%
10. Patients must have the ability to swallow and retain oral medication
11. Toxicities from prior therapy greater than CTCAE Grade 1 have resolved with the exception of alopecia. Patients with Grade ≤ 2 neuropathy are eligible.
12. Male patients with female partners of child-bearing potential must be willing to use two forms of acceptable contraception, including one barrier method, during their participation in this study and for 6 months after stopping study treatment with olaparib and/or AZD5153. Female partners of child-bearing potential of male patients must use at least one of the two forms of acceptable contraception.

    * Male patients must agree to refrain from donating sperm during their participation in the study and until 6 months after the last treatment with olaparib and/or AZD5153.
    * Male patients will be counselled about the effects of the drug on their fertility and the utility of freezing their sperm samples prior to the start of the study should they wish to father children while on AZD5153 or during the 6 months after stopping AZD5153.
13. Female patients must use two highly effective contraceptive measures. All methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by a male sexual partner for intercourse. Female patients must not be breast-feeding and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment.
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.

Additional Inclusion Criteria Specific for Monotherapy Dose Escalation:

1. Patients with histological or cytological confirmation of a malignant solid tumor (locally advanced or metastatic) or lymphoma (any histology) that is refractory to standard therapy(ies) or for which no standard therapy(ies) exists.

   - Patients with a malignant solid tumor must have at least 1 lesion that can be accurately measured at baseline by computed tomography (CT) scan according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria (Eisenhauer et al. 2009) and is suitable for repeated measurement.
2. Patients with lymphoma must have documented analysis of bone marrow infiltration from biopsy carried out < 3 months of enrollment, or be able to undergo a new bone marrow biopsy if such procedure was performed > 3 months prior to enrollment.

   - Patients with a lymphoma must have at least 1 lesion that can be accurately assessed at baseline by CT or CT and positron emission tomography (PET) according to the Cheson criteria (Cheson et al 2007 and is suitable for repeated assessment.
3. Patient must agree to the collection of formalin fixed paraffin-embedded (FFPE) blocks or slides from archival diagnostic histology samples, or a fresh pre-treatment biopsy will be accepted.

Additional Inclusion Criteria specific for MTD monotherapy expansion and olaparib combination dose escalation:

1. Patients with the following histologies that have at least 1 lesion that can be accurately assessed at baseline by CT scan according to RECIST v1.1 criteria (Eisenhauer et al. 2009) and is suitable for repeated assessment:

   1. Histologically or cytologically confirmed platinum-resistant OR platinum-refractory HGSO, fallopian, or primary peritoneal cancer in the relapsed setting. Platinum-resistant disease is defined by progression within 6 months following the last administered platinum-based regimen. Platinum-refractory disease is defined by lack of at least a partial response while on platinum-containing regimens.
   2. Triple-negative breast cancer (TNBC) that is refractory to standard therapy(ies) or for which no standard therapy(ies) exists
   3. Refractory metastatic castrate-resistant prostate cancer (mCPRC)
   4. Pancreatic ductal adenocarcinoma (PDAC) with progression on standard treament
2. Patients will be allowed on study regardless of their BRCA mutational status. Information about their BRCA mutational status or other HRD gene mutational status must be collected if patients have been tested as part of their standard of care.
3. Previous response to olaparib or other PARPi is not required
4. Patients must have at least 1 site of disease amenable to biopsy at screening, and must be a candidate for tumor biopsy. Patients must be willing to undergo a new tumor biopsy during screening. An on-treatment tumor biopsy will be mandatory in the olaparib combination dose escalation portion of this study, and optional from consenting patients in the monotherapy expansion at MTD.
5. For the olaparib combination portion of this study, patients are required to have hemoglobin ≥10 g/dL at study entry.

Exclusion Criteria:

1. Patients who have been treated with most recent chemotherapy, radiotherapy, hormonal therapy, immunotherapy or investigational drugs within 21 days or 5 half-lives (whichever is shorter) from enrollment.
2. Minimum wash-out period for previous PARPi therapy is at least 14 days or 5 half-lives whichever is shorter, or until toxicity from previous PARPi therapy has fully recovered.
3. Patient received more than 5 prior lines of treatment for an advanced solid tumor (including HGSO cancer, TNBC, mCRPC, or PDAC). Patients with lymphoma will be able to enroll without a restriction in the number of previous therapies received, if they otherwise meet eligibility criteria.
4. Major surgery (excluding placement of vascular access) ≤ 21 days from the beginning of enrollment or minor surgical procedures ≤ 7 days. No waiting is required following implantable port and catheter placement.
5. Patient is unable to swallow oral medications or has a gastrointestinal disorder (e.g., malabsorption) that would jeopardize intestinal absorption of AZD5153 and olaparib.
6. Treatment with any of the following:

   * Patient has had prescription or non-prescription drugs or other products known to be strong or moderate inhibitors/inducers of CYP3A4/5, or CYP3A4/5 sensitive substrates or substrates with a narrow therapeutic range, which cannot be discontinued 2 weeks prior to the first day of dosing and withheld throughout the study until 2 weeks after the last dose of AZD5153 and/or olaparib.
   * Drugs that are sensitive substrates of the transporters P-gp, UGT1A1, BCRP, OATP1B1, OAT3, OCT1, OCT2, MATE1 and MATE2K.
   * Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, kava, ephedra (ma huang), ginkgo biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Patients should stop using these herbal medications 14 days prior to the first dose of AZD5153 and/or olaparib.
   * Drugs known to prolong QT interval or induce Torsades de Pointes.
7. Refractory nausea and vomiting, previous significant bowel resection that would preclude adequate absorption of study drug and chronic gastrointestinal disease including active or prior documented inflammatory bowel disease.
8. Patient has a history of tuberculosis.
9. Patients receiving a live attenuated vaccine ≤28 days before the first dose of study drug.
10. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
11. A diagnosis of MDS or secondary AML (for olaparib combination dose escalation only)
12. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or other comorbidity that renders the patient unsuitable for participation in the study. Screening for chronic conditions is not required.
13. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTcF) >450 msec obtained from 3 electrocardiograms (ECGs).
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third degree heart block.
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age.
14. History of hypersensitivity to active or inactive excipients of AZD5153 and/or olaparib or drugs with a similar chemical structure or class to AZD5153 and/or olaparib.
15. Patients with non-Hodgkin lymphoma (NHL) at high risk for developing tumor lysis syndrome are not eligible for the monotherapy dose escalation part of this study.
16. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
17. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT). | From the first dose of study treatment up to last day of cycle 1 (21 days)
  DLTs will be determined from monitoring adverse events (AEs), and abnormal laboratory tests (clinical chemistry, hematology, and urinalysis), physical examinations, vital signs (blood pressure and pulse), and electrocardiogram (ECG).

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood and plasma will be determined (Cmax will be derived).
The urine concentration of AZD5153 and its co-former (if appropriate). | Urine will be collected pre-dose (spot sample), and volumetrically from 0-6, 6-12, 12-24 hours on Day 1 and Day 15 of Cycle 1.
  Total urine volume will be measured for each interval and urine concentration of AZD5153 will be determined. A sample for the determination of 1β-hydroxy deoxycholic acid will be taken from the total urine collection at each scheduled time interval.
The effect of AZD 5153 on QTc interval. | ECGs will be performed at prespecified time points on Days 1 and 2 and 15 and 16 of Cycle 1.
  Triplicate 12-lead ECGs will be taken at screening and at prespecified times on Cycle 1 Days 1 and 2 and Days 15 and 16.
Antitumor activity of AZD5153 in patients by assessing the disease control rate (DCR). | Up to 1 year
  Investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for solid tumors or the 2007 Revised Response Criteria for Malignant Lymphoma criteria for lymphoma will be applied.
  The preliminary anti-tumor activity of AZD5153 in patients with ovarian carcinoma will be evaluated.
Antitumor activity of AZD5153 in patients by assessing progression free survival (PFS). | Up to 1 year
  Investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for solid tumors or the 2007 Revised Response Criteria for Malignant Lymphoma criteria for lymphoma will be applied.
Antitumor activity of AZD5153 in patients by assessing overall response rate (ORR). | Up to 1 year
  Investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for solid tumors or the 2007 Revised Response Criteria for Malignant Lymphoma criteria for lymphoma will be applied.
  The preliminary anti-tumor activity of AZD5153 in patients with ovarian carcinoma will be evaluated.
Antitumor activity of AZD5153 in patients by assessing duration of response (DoR). | Up to 1 year
  Investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for solid tumors or the 2007 Revised Response Criteria for Malignant Lymphoma criteria for lymphoma will be applied.
  The preliminary anti-tumor activity of AZD5153 in patients with ovarian carcinoma will be evaluated.
Area under the plasma concentration versus time curve (AUC). | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood will be determined. Area under the curve is the integral of the concentration-time curve. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration. The area under the curve is dependent on the rate of elimination of the drug from the body and the dose administered.
Time to reach peak plasma concentration (tmax). | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood will be determined. Tmax is the time required after administration for the drug to reach its peak plasma concentration.
Elimination half-lfe (t1/2). | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood will be determined. Elimination half-life (t1/2) is the time required for the concentration of the drug to reach half of its original value.
Volume of distribution (Vd). | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood will be determined. Volume of distribution (Vd) is the apparent volume in which a drug is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
Clearance (CL). | Samples for single dose PK will be collected at prespecified time points on Day 1, Cycle 1 pre-dose on Day 2. Multiple-dose PK will be assessed from samples taken on Days 15 and 16 of Cycle 1.
  The concentration of AZD5153 and its co-former in blood will be determined. Clearance (CL) is the volume of plasma cleared of the drug per unit time.

CONTACTS AND LOCATIONS:
Overall Officials: Erika P Hamilton, MD, Principal Investigator — Sarah Cannon
Locations (4):
- United States (3):
  - Research Site, Sarasota, Florida
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
- Research Site, Toronto, CA, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home